CLINICAL TRIAL: NCT07088367
Title: The Effect of Virtual Reality Meditation on Anxiety Management in Cancer Patients Receiving Chemotherapy: A Randomized Controlled Study
Brief Title: Virtual Reality Meditation on Anxiety in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulbeyaz Can, Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-126
Record Dates: First submitted 2025-06-12; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Cancer
Keywords: cancer; anxiety
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality meditation group (Experimental): Participants in this group will use a virtual reality (VR) headset to complete a 10-minute meditation session on three consecutive days. A different meditation video will be used each day, and sessions will be held between 10:00 AM and 12:00 PM. The meditation sessions are provided through the "MediboothVR" application. This app is the first immersive virtual reality meditation tool developed in Türkiye and supports the Turkish language.
  In MediboothVR, participants experience a 360-degree guided meditation in a virtual environment. Each video starts with a short environmental scene, followed by a visual journey to a meditation space where a guiding silhouette appears and leads the participant through the session. Each session lasts approximately 10 minutes.
  Interventions: Behavioral: Virtual reality meditation
- Virtual Reality Video Group (Active Comparator): This group will use a VR headset on three consecutive days between 10:00 AM and 12:00 PM. Instead of meditation, participants will watch 360-degree nature videos. A different video (10 minute) will be shown each day. The purpose is to create a calming, immersive experience without guided meditation.
  Interventions: Behavioral: Virtual Reality Videos
- Control Group (No Intervention): Participants in the control group will receive standard nursing care without any VR intervention.

INTERVENTIONS:
Behavioral: Virtual reality meditation — This intervention involves immersive virtual reality (VR)-based guided meditation sessions using MediboothVR, the first Turkish-language supported virtual reality meditation application developed in Türkiye. It is distinct from other VR interventions in the following ways:
  Cultural and language adaptation: MediboothVR is fully available in Turkish, providing culturally relevant audio-guided content. This makes it more accessible and emotionally resonant for Turkish-speaking participants, unlike many VR applications designed in other languages.
  Duration and consistency: The intervention is delivered over three consecutive days, with a different video used each day, each lasting approximately 10 minutes.
  Technical delivery: The application is used exclusively via VR headsets, creating a fully immersive experience that eliminates visual and auditory distractions from the hospital environment.
  Arms: Virtual reality meditation group
Behavioral: Virtual Reality Videos — This intervention involves the use of a virtual reality headset to present immersive 360-degree calming nature videos to participants. It is distinct from other video- or relaxation-based interventions in several key ways:
  Delivery via VR headset: Unlike standard video-based relaxation interventions presented on screens or tablets, this method delivers video content in a fully immersive virtual reality environment, which blocks out external visual and auditory stimuli from the unit.
  Non-guided and passive exposure: The video group receives no audio-guided instruction or meditation scripting, making it a purely visual and passive exposure intervention.
  Cultural relevance and visual neutrality: The nature videos are non-verbal, visually neutral, and free of religious, symbolic, or emotionally provocative imagery, allowing them to be suitable for a diverse patient population.
  Arms: Virtual Reality Video Group

SUMMARY:
The main questions this study aims to answer are:

Does VR meditation, delivered through virtual reality glasses and the MediboothVR application, effectively reduce anxiety in cancer patients during chemotherapy?

Is there a meaningful difference in anxiety reduction between the VR intervention groups and the control group?

Researchers will compare two intervention groups using VR glasses-one with guided meditation and one with calming video content-to a control group receiving standard care, to see if there are differences in anxiety levels.

Participants will:

Be randomly assigned to one of three groups

Attend their scheduled chemotherapy sessions

Depending on group assignment, either:

Use VR glasses with the MediboothVR meditation app for 10 minutes daily

Use VR glasses to watch calming 360-degree nature videos for 10 minutes daily

Receive standard care with no VR use

All participants will complete anxiety questionnaires and have their vital signs recorded before and after each session.

DETAILED DESCRIPTION:
This clinical trial includes three parallel groups: a VR meditation group, a VR video group, and a control group.

Participants in the VR meditation group will receive a 10-minute virtual reality (VR) guided meditation session on three consecutive days, between 10:00 AM and 12:00 PM. The sessions will be delivered using virtual reality glasses and the MediboothVR application. A different meditation video will be used each day.

The MediboothVR application is the first immersive virtual reality meditation app developed in Türkiye and is also the first to support the Turkish language. It provides audio-guided meditation in a 360-degree artificial environment through virtual reality glasses. Each meditation video lasts approximately 10 minutes. Sessions begin with a short period for environmental observation, followed by a journey sequence that transports the user to a dedicated meditation area. A silhouette then appears and delivers the guided meditation experience through structured audio.

Participants in the VR video group will also use virtual reality glasses for 10 minutes each day, over three consecutive days, during the same time frame. Instead of meditation, they will watch 360-degree calming nature videos. A different video will be shown each day to support relaxation through immersive visual content.

These videos were selected to promote relaxation and included high-definition panoramic visuals such as forests, oceans, waterfalls, and mountain landscapes. Each day, a different video was used to maintain novelty and reduce visual fatigue. Although no verbal instructions were provided, the rich sensory environment was designed to offer a passive but calming distraction from the clinical setting.

Participants in the control group will receive standard nursing care without any VR-based intervention. After data collection is completed, participants in the control group will be offered the opportunity to experience the VR content, but their responses will not be included in the study analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* Sufficient communication ability to respond to study questions,
* Receiving outpatient treatment for at least three consecutive days with a confirmed cancer diagnosis,
* Scoring 40 or above on the State Anxiety Inventory (STAI-S), indicating moderate or higher anxiety levels,
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Inability to speak or understand Turkish,
* Being under contact isolation precautions,
* Presence of active eye discharge or visual impairment,
* History of seizures, epilepsy, or hypersensitivity to flashing lights,
* History of vertigo or motion sickness,
* Experiencing active nausea or vomiting,
* Having wounds or dressings on the head or face that interfere with the use of a VR headset,
* Hearing impairment,
* Hypersensitivity of the face or scalp to light pressure,
* Diagnosis of psychiatric conditions that may affect participation (e.g., schizophrenia, severe psychosis),
* Diagnosis of recurrent or relapsed cancer,
* Scoring below 40 on the State Anxiety Inventory,
* Previous use of virtual reality applications,
* Prior experience with meditation practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
State Anxiety | Immediately Before and after each intervention session, on Day 1, Day 2, and Day 3 (total of 6 measurement points)
  Change in State Anxiety Score
  Anxiety levels will be measured using the State Anxiety subscale of the State-Trait Anxiety Inventory (STAI-S), a validated self-report tool.
  The STAI-S consists of 20 items. Each item is rated on a 4-point Likert scale (1 = Not at all, 4 = Very much so). Total scores range from 20 to 80, with higher scores indicating greater anxiety.
  Participants will complete the STAI-S before and after each VR session (or standard care, in the control group) on three consecutive days. This outcome will evaluate daily changes in state anxiety levels, and whether the intervention (VR meditation or VR video) leads to a significant reduction in anxiety compared to control.

SECONDARY OUTCOMES:
Trait Anxiety | Day 1 (baseline, before the first intervention),Day 3 (after the last intervention session), andDay 30 (follow-up assessment)
  Trait anxiety will be measured using the Trait Anxiety subscale of the State-Trait Anxiety Inventory (STAI-T), a validated self-report instrument.
  The STAI-T consists of 20 items rated on a 4-point Likert scale (1 = Almost never, 4 = Almost always). Total scores range from 20 to 80, where higher scores indicate higher levels of trait (long-term) anxiety.
  This outcome will assess changes in trait anxiety scores across three time points (baseline, post-intervention, and follow-up) to evaluate the immediate and sustained effects of virtual reality-based interventions compared to standard care. A reduction in scores will indicate a positive effect on long-term anxiety regulation.
Virtual Reality Sickness | Immediately after each VR session on Day 1, Day 2, and Day 3
  Virtual reality-induced discomfort will be assessed using the Virtual Reality Sickness Questionnaire (VRSQ), a standardized and validated instrument designed to measure symptoms such as dizziness, nausea, eye strain, and general discomfort during or after VR use.
  The VRSQ consists of multiple items scored on a Likert-type scale. Higher total scores indicate greater levels of VR-induced discomfort.
  This outcome will help evaluate the tolerability and usability of VR-based interventions in cancer patients receiving chemotherapy. It will also identify whether repeated exposure over three days influences the presence or intensity of VR sickness symptoms.
  Note: This assessment is only applied to participants in the virtual reality meditation and VR video groups, and is not administered to the control group.
Participant Satisfaction with VR Intervention | Immediately after each VR session on Day 1, Day 2, and Day 3
  Satisfaction with the virtual reality experience will be evaluated using a single-item visual analog scale ranging from 0 to 10, where:
  0 = Not satisfied at all
  10 = Extremely satisfied
  This outcome will assess how participants perceived the comfort, usefulness, and overall satisfaction with the VR-based meditation or video intervention. Only participants in the intervention groups (VR meditation and VR video) will complete this measure.
Participant's Heart Rate | Immediately before and after each VR session on Day 1, Day 2, and Day 3.
  Vital signs will be measured immediately before and after each intervention session to assess the short-term physiological effects of the virtual reality experience. The following parameters will be recorded:
  Heart rate (per minute)
  Changes in these vital signs will be analyzed to determine whether the VR meditation or VR video sessions have any immediate impact on participants' physiological responses. The control group's measurements were taken at time points corresponding to those used in the intervention groups (e.g., 10 minutes after start for pre-test, 25th minute for post-test).
Participant's Respiratory Rate | Immediately before and after each VR session on Day 1, Day 2, and Day 3.
  Vital signs will be measured immediately before and after each intervention session to assess the short-term physiological effects of the virtual reality experience. The following parameters will be recorded:
  Respiratory rate (breaths per minute)
  Changes in these vital signs will be analyzed to determine whether the VR meditation or VR video sessions have any immediate impact on participants' physiological responses. The control group's measurements were taken at time points corresponding to those used in the intervention groups (e.g., 10 minutes after start for pre-test, 25th minute for post-test).
Participant's Blood Pressure | Immediately before and after each VR session on Day 1, Day 2, and Day 3.
  Vital signs will be measured immediately before and after each intervention session to assess the short-term physiological effects of the virtual reality experience. The following parameters will be recorded:
  Blood pressure (mmHg)
  Changes in these vital signs will be analyzed to determine whether the VR meditation or VR video sessions have any immediate impact on participants' physiological responses. The control group's measurements were taken at time points corresponding to those used in the intervention groups (e.g., 10 minutes after start for pre-test, 25th minute for post-test).
Participant's Oxygen Saturation | Immediately before and after each VR session on Day 1, Day 2, and Day 3.
  Vital signs will be measured immediately before and after each intervention session to assess the short-term physiological effects of the virtual reality experience. The following parameters will be recorded:
  Oxygen saturation (SpO₂, %)
  Changes in these vital signs will be analyzed to determine whether the VR meditation or VR video sessions have any immediate impact on participants' physiological responses. The control group's measurements were taken at time points corresponding to those used in the intervention groups (e.g., 10 minutes after start for pre-test, 25th minute for post-test).

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Results will be reported at the group level in scientific publications.

REFERENCES:
- [Background] Uslu A, Arslan S. The Effect of Using Virtual Reality Glasses on Anxiety and Fatigue in Women with Breast Cancer Receiving Adjuvant Chemotherapy: A Pretest-Posttest Randomized Controlled Study. Semin Oncol Nurs. 2023 Oct;39(5):151503. doi: 10.1016/j.soncn.2023.151503. Epub 2023 Sep 22. PMID 37741768
- [Background] Franklin, D. M., Silvestro, C., Carrillo, R. A., Yang, Y., Annadurai, D., Ganesan, S., Vasantham, D. S. J., Mettu, S., Patel, M., Patil, M. S., & Akurathi, N. D. (2023). The impact of meditation aided by VR technology as an emerging therapeutic to ease cancer related anxiety, stress, and fatigue. Frontiers in Virtual Reality, 4(July), 1-12. https://doi.org/10.3389/frvir.2023.1195196
- [Background] Wu Y, Wang N, Zhang H, Sun X, Wang Y, Zhang Y. Effectiveness of Virtual Reality in Symptom Management of Cancer Patients: A Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2023 May;65(5):e467-e482. doi: 10.1016/j.jpainsymman.2023.01.023. Epub 2023 Feb 8. PMID 36758907
- [Background] Chow H, Hon J, Chua W, Chuan A. Effect of Virtual Reality Therapy in Reducing Pain and Anxiety for Cancer-Related Medical Procedures: A Systematic Narrative Review. J Pain Symptom Manage. 2021 Feb;61(2):384-394. doi: 10.1016/j.jpainsymman.2020.08.016. Epub 2020 Aug 19. PMID 32822755
- See also: MediboothVR application — https://www.mediboothvr.com/
- See also: Nature Video: Virture Forest Walk — https://www.youtube.com/watch?app=desktop&v=Ba7f8xNKfVY&t=1s
- See also: Nature Video: Wetland Marsh Bird Sounds — https://www.youtube.com/watch?v=CorMkB9EHo0&t=1274s
- See also: Nature Video: Stones of the Skagit River — https://www.youtube.com/watch?v=mBWj443FNGs&t=2519s